CLINICAL TRIAL: NCT03398720
Title: A Two-Part, Phase 1, Open-Label, Multicenter, Non-Randomized, Dose Escalation/Expansion Study to Evaluate the Safety and Tolerability of HTI-1066 in Subjects With Advanced Solid Tumors
Brief Title: Safety and Tolerability of HTI-1066 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTI-1066-101
Record Dates: First submitted 2017-12-26; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): One participant will receive HTI-1066 at the starting dose.
  Interventions: Drug: HTI-1066 dose level 1
- Cohort 2 (Experimental): Participants will receive HTI-1066 at dose level 2.
  Interventions: Drug: HTI-1066 dose level 2
- Cohort 3 (Experimental): Participants will receive HTI-1066 at dose level 3.
  Interventions: Drug: HTI-1066 dose level 3
- Cohort 4 (Experimental): Participants will receive HTI-1066 at dose level 4.
  Interventions: Drug: HTI-1066 dose level 4

INTERVENTIONS:
Drug: HTI-1066 dose level 1 — Starting dose level
  Arms: Cohort 1
Drug: HTI-1066 dose level 2 — 2nd dose level
  Arms: Cohort 2
Drug: HTI-1066 dose level 3 — 3rd dose level
  Arms: Cohort 3
Drug: HTI-1066 dose level 4 — 4th dose level
  Arms: Cohort 4

SUMMARY:
HTI-1066 is a novel ADC being developed for the treatment of cancers in patients with overexpression of c-Met. This 2-part, Phase 1 study evaluates the safety the tolerability of HTI-1066 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a 2-part dose escalation and dose expansion study. Dose escalation uses a modified "3+3" design and continues until a maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) is identified. In part 2, subjects with selected tumor types will be enrolled at the MTD or RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Subject must have an advanced solid tumor
3. ECOG Performance Status of 0 or 1
4. Life expectancy ≥12 weeks
5. Adequate laboratory parameters
6. Female subjects agree not to be pregnant or lactating from beginning of the study screening until 4 months after receiving the last treatment; Male and female subjects and their sexual partners are willing and able to employ a highly effective method of birth control/contraception.
7. Willing and able to comply with clinic visits and study-related procedures
8. Provide signed informed consent

Exclusion Criteria:

1. Hypersensitivity to HTI-1066 or sensitivity to humanized monoclonal antibody products
2. Any concurrent therapy for cancer, radiation, or surgery within 4 weeks, except for minor palliative intent (this is to be discussed with sponsor)
3. Any concurrent use of anti-infective, anti-fungal, or anti-viral agent (exceptions are to be approved by the sponsor)
4. Any other prohibited or restricted medication as described in the study protocol.
5. Investigational therapy administered <5 half-lives before the first dose of HTI-1066
6. Any anticancer therapy administered <5 half-lives before first dose of HTI-1066; any prior immune-oncology products administered within 4 weeks or 5 half-lives before the first dose of HTI-1066 as described above; or surgery or radiotherapy administered within 4 weeks before the first dose of HTI-1066.
7. Active CNS metastases.
8. Cardiac disease (NYHA classes II-IV) including myocardial infarction within 6 months before enrollment, or unstable angina, congestive heart failure, or cardiac arrhythmia requiring treatment.
9. History or presence of an abnormal ECG, ECHO, or MUGA that is clinically meaningful.
10. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or any active systemic viral infection requiring therapy (e.g., hepatitis B or C)
11. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare or ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
12. Active infection or an unexplained fever >38.5°C during Screening or on the first scheduled day of dosing.
13. Unresolved toxicities from previous anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-31 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 2 year
  Number of participants with AEs and SAEs
Dose-limiting toxicity (DLT) | Up to 2 years
  Number of participants with DLTs

SECONDARY OUTCOMES:
AUC | Up to 1 year
  Area under the curve
Cmax | Up to 1 year
  Peak concentration at Tmax
Anti-drug antibodies | Up to 2 year
Objective response rate | Up to 2 years
Progression-free survival (PFS) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Sarah Cannon - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No